CLINICAL TRIAL: NCT03978962
Title: Performance and Safety of the Resorbable Collagen Membrane "Ez Cure" in Guided Tissue Regeneration and Guided Bone Regeneration Procedures
Brief Title: Performance and Safety of the Resorbable Collagen Membrane "Ez Cure"
Status: Completed | Type: Observational
Sponsor: Biomatlante (Industry)
Collaborators: Atlanstat (Industry)
Responsible Party: Sponsor
Other Study IDs: RE-DT04-18A; 2018-A03202-53 (Other: ANSM)
Record Dates: First submitted 2019-05-07; First posted 2019-06-07 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Oral Bone Defect; Maxillofacial Bone Defect; Periodontal Bone Loss; Alveolar Bone Loss
Keywords: Periodontal defects; Alveolar bone preservation; Collagen membrane; Mucosa healing
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Guided Tissue Regeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study population: Patients subjects to a Guided Tissue Regeneration or Guided Bone Regeneration procedure
  Interventions: Device: Guided Tissue Regeneration

INTERVENTIONS:
Device: Guided Tissue Regeneration — Covering oral-maxillofacial or a periodontal defects with the Resorbable Collagen Membrane in order to avoid epithelial cell infiltration and to promote periodontal tissues healing.
  Covering alveolar bone defects after tooth-teeth extraction.
  Other Names: Guided Bone Regeneration

SUMMARY:
The evaluation of the clinical data has demonstrated the conformity of the Resorbable Collagen Membrane (RCM), EZ CureTM, with the relevant essential requirements for its use in periodontal applications. The RCM is intended for Guided Tissue Regeneration (GTR) and Guided Bone Regeneration (GBR) procedures. It acts as a barrier against the migration of epithelial cells within the bone defect (performance) and thus complies with several surgical indications in the treatment of maxillofacial bone defects. It has been concluded that the risks associated with the use of this device are acceptable when weighted against the benefits to the patients.

In order to improve the clinical data on the RCM, the manufacturer, Biomatlante, decided to assess that the performance and safety of the device are maintained until the reaching of its intended use. In this objective, the goal of this study will be to observe the following parameters:

1. Tissue regeneration (mucosa health on the site of implantation)
2. Safety (report of any adverse event)
3. Radiographic analysis of periodontal tissues

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged from 18 to 70
* Periodontal defects (e.g. cyst, bone tumour, crest augmentation...)
* Aleveolar bone defect after tooth (teeth) extraction
* Non opposition form (consent of the patient)
* Patients affiliated to the French social security
* Patients not under guardianship or judicial protection

Exclusion Criteria:

* Pregnancy of breastfeeding women
* Severe smoker (>10 cigarettes per day)
* Acute infections
* Allergies to the material (if an allergy of any kind is suspected, adequate exams must be carried out in advance)
* Refusal of the patient to adhere to surgical follow-up and to the limit in activity level
* Fever and/or local inflammation
* HIV positive known
* History of uncontrolled diabetes (untreated or not stabilized by treatment)
* History of treatments for previous corticosteroids, long-term (more than 6 months) and interrupted for less than 3 months
* History of chemotherapy in progress or during the last three months
* History of cervico-facial radiotherapy
* History of bone disease with disorders of blood circulation which is defined as Akbers-Schönberg disease or Paget's disease
* Known severe hyperparathyroïdism
* History of severe immune deficiency

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The group will be selected in the entire population of the dental care center
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2020-08-26 (Actual); Study Completion 2020-08-26 (Actual)

PRIMARY OUTCOMES:
Change of the patient's mucosa health in terms of swelling, wound closure and colour of the implantation site (visual inspection) | 1 week post-surgery (+/-2 days) / 2 weeks post-surgery (+/-2 days) / 12 weeks post-surgery (+/-1 week)
  Observation of the change of the mucosa health in terms of swelling, wound closure and colour of the implantation site. It reflects the performance of the Resorbable Collagen Membrane

SECONDARY OUTCOMES:
Number and precise description of any adverse event during the follow-up | From screening visit through visit at 12 weeks
  Record and description of any adverse event during the follow-up that reflects the safety of the Resorbable Collagen Membrane
Percentage of bone reconstruction in the treated bone defect by a radiographic examination | Before surgery and 12 weeks post-surgery (+/-1 week)
  Comparison of the radiographies recorded before surgery and at the last follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Saïd Kimakhe, PhD, DDS, Principal Investigator — Centre Hospitalo-Universitaire de Nantes; Saïd Kimakhe, Phd, DDS, Principal Investigator — Cabinet privé; Guy Daculsi, PhD, Study Director — Biomatlante
Locations (2):
- France (2):
  - Centre de soins dentaires - Centre Hospitalo-Universitaire de Nantes, Nantes
  - Cabinet privé du Dr. S. Kimakhe, Nantes

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/62/NCT03978962/Prot_SAP_000.pdf